CLINICAL TRIAL: NCT05671913
Title: Effects of Opioid Requirements With Scheduled Intranasal Ketamine During Admission for Traumatic Pain
Brief Title: Scheduled Intranasal Ketamine
Acronym: SINK
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding not acquired to run the study.
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SH Briggs IN Ketamine
Record Dates: First submitted 2022-07-13; First posted 2023-01-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pain; Trauma
MeSH Terms: conditions — Pain; Wounds and Injuries | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Intranasal Ketamine
  Interventions: Drug: Ketamine
- Control (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Treatment arm
  Arms: Treatment
Drug: Placebo — Control arm
  Arms: Control

SUMMARY:
The purpose of this research is to determine if scheduled intranasal ketamine effects opioid requirements in adult trauma patients with moderate to severe pain in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient between aged 18-80 years, present following a traumatic incident, rate pain > 5 on the numeric rating scale (NSR), and require admission to the hospital.

Exclusion Criteria:

* - Patients that arrive at facility intubated
* Patients that received Ketamine in the field
* Patients less than 18 years old or greater than 80 years
* Pregnant or breast-feeding females
* Hemodynamic instability defined as need for vasoactive drugs or Systolic blood pressure >180
* Weight less than 80 pounds or greater than 300 pounds
* Glasgow Coma Scale less than 15
* Current acute head injury resulting in unconsciousness
* Current or history of eye injury
* Current or history of seizures
* Facial or nasal fractures that require nasal precautions
* Current or history of intracranial hypertension
* History of Schizophrenia
* BAC (Blood Alcohol Content) greater than 0.08
* Current alcohol abuse
* Current drug abuse or positive drug screen
* Chronic pain or patients on pain contracts
* Inability to assess pain intensity
* Contraindications or allergies to the treatment
* Patients with hepatic insufficiency
* Prisoners
* Nursing home residents
* Urine drug screen positive for illicit drugs or medications not on their home medication list.
* BAC > 0.08
* Positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Morphine Equivalents (TME) throughout hospitalization | 72 hours
  Total Morphine Equivalents is a standardized way of measuring opioids that patients receive over time. This will be calculated by a member of the research study team utilizing a standardized formula under pharmacies direction. The Medication Administration Record (MAR) will be reviewed to gather administered doses of opioids throughout the participants hospital stay.

IPD SHARING:
Plan to Share IPD: No